CLINICAL TRIAL: NCT06926959
Title: Tricuspid RegurgitAtion rIsk modeL Study (TRAIL Study)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Hospital of Guangdong Medical University (Other); Second Affiliated Hospital of Shantou University Medical College (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Jieyang People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, Sun Yat-sen University
Other Study IDs: TRAIL study
Record Dates: First submitted 2025-03-24; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid Regurgitation; all-cause mortality; risk factor; prediction model
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a multicenter cohort study including patients diagnosed with tricuspid regurgitation during hospitalization. The primary outcome of the study is all-cause death, and the secondary outcome is cardiovascular events. The prognostic risk factors of patients with tricuspid regurgitation are evaluated, and the prognostic models are constructed through the follow-up observation.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 yrs.
* Patients diagnosed with tricuspid regurgitation during hospitalization.

Exclusion Criteria:

* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with tricuspid regurgitation (TR) during hospitalization were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-06-15 (Actual); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | Through study completion, an average of 5 years
  Death due to any cause after enrollment

SECONDARY OUTCOMES:
Cardiovascular death | Through study completion, an average of 5 years
  Death caused by cardiac causes
Heart Failure Hospitalization | Through study completion, an average of 5 years
  Hospitalization with the primary reason for admission as acute decompensated HF and administration of intravenous or mechanical heart failure therapies.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Sun Yat-sen Univerity, Guangzhou, Guangdong
  - Third Affiliated Hospital, Sun Yat-Sun University,, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Eighth Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong